CLINICAL TRIAL: NCT04170478
Title: Transperineal Laser Ablation for Focal Prostate Cancer: Safety and Ablative Efficacy Evaluation Using Postradical Prostatectomy Histological Analysis
Brief Title: Transperineal Laser Ablation for Focal Treatment of Prostate Cancer
Acronym: TPLA for PCa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Elesta S.R.L. (Industry); Amsterdam UMC, location VUmc (Other); The Netherlands Cancer Institute (Other)
Responsible Party: Principal Investigator, Prof.dr. H.P. Beerlage, Head of Urology department, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019_161; NL69903.018.19 (Other: Toetsingonline)
Record Dates: First submitted 2019-10-30; First posted 2019-11-20 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Prostate Cancer; Focal Laser Ablation; Transperineal Laser Ablation
Keywords: Prostate Cancer; Transperineal laser ablation; Prostate neoplasma; Focal laser ablation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Echolaser X4 system — Transperineal laser ablation

SUMMARY:
Rationale: Prostate cancer (PCa) is the second cause of cancer-related deaths for men. The standard surgical treatment for localised prostate cancer is radical prostatectomy. Possible side effects of this treatment are incontinence and erectile dysfunction and this is related to the whole-gland resection. A focal treatment with fewer side effects is desired for patients with only a small focus of PCa. For this purpose, focal laser ablation is feasible. Current focal laser ablation techniques use a single fibre setup with the need for fibre replacement revisualisation of the tumour side accordingly. This leads to a long treatment duration.

The Echolaser® system is a laser ablation system with four simultaneously operating laser sources. This provides a potential larger treatment area, without the need for fibre replacement.

This makes the system advantageous for focal laser ablation of prostate cancer, especially since it can be applied under local anaesthesia.

This pilot study aims to evaluate histological ablative efficacy on radical prostatectomy specimens following TPLA, feasibility and safety using a (multi)fibre setup in men with localized prostate cancer. The investigators hypothesize that TPLA will show adequate histological ablative efficacy and will be feasible and safe.

ELIGIBILITY:
Inclusion Criteria:

* Male
* ≥40 years of age
* Histopathological confirmed organ-confined prostate cancer
* Indication for a radical prostatectomy
* Prostate volume ≥40 mL
* Ability of the patient to stop anticoagulant therapy prior to TPLA according to standard hospital pre-operative protocol
* Signed informed consent

Exclusion Criteria:

* Refusal of participation or clinically ineligible for treatment under local anaesthesia
* Prior or concurrent treatment for prostate cancer
* Other conditions / status

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Ablative efficacy of transperineal laser ablation determined by size of the ablation zone in histopathology, which is measured by absence of vital prostatic cells, compared to the size measured on imaging (CEUS/MRI) during and after treatment | 30 days following TPLA treatment
  Histological ablative efficacy is assessed on histopathological analysis of the prostatic tissue after radical prostatectomy by means of the absence of vital cells in the treated prostate zone

SECONDARY OUTCOMES:
Safety is assessed by device and procedural adverse events using the CTCAEv5.0 until radical prostatectomy and feasibility is determined by procedural success of the TPLA treatment. | 30 days following TPLA treatment
  Safety is assessed by device and procedural adverse events using the CTCAE v5.0 until radical prostatectomy. TPLA is definitely safe when ≤10% of patients experience major adverse events, defined as grade 3 or higher. Technical feasibility is determined by procedural success of the TPLA treatment.
  TPLA is definitely feasible when ≥90% of procedures is performed successfully without any problems regarding needle placement, fibre introduction or device malfunctioning.
Size of ablation zone | 30 days following TPLA treatment
  Determination of the size of the ablated area
Observation of tissue changes seen on imaging during and after treatment compared to histopathology | 30 days following TPLA treatment
  Ablation zone volumes are measured using CEUS and mpMRI and these are used to determine ablation zone compared to histopathological changes. Visual changes are identified and described.
Functional outcomes measured using PROMs (VAS, IPSS, IIEF-15, EPIC) | 30 days following TPLA treatment
  Determination of short-term functional outcomes following TPLA treatment

CONTACTS AND LOCATIONS:
Overall Officials: J R Oddens, MD, PhD, Principal Investigator — Urologist
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided